CLINICAL TRIAL: NCT05580393
Title: Molecular Characterization of Blastocystis Isolates From Human by Restriction Fragment Length Polymorphism (RFLP) Analysis in Sohag Governorate
Brief Title: Molecular Characterization of Blastocystis Isolates From Human by Restriction Fragment Length Polymorphism (RFLP) Analysis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shimaa Refaey Mohamed Abd-Elal, Assistant Lecturer, Sohag University
Other Study IDs: Soh-Med-22-10-16
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Blastocystis Infections
Keywords: Blastocystis; colorectal cancer; irritable bowel syndrome
MeSH Terms: conditions — Blastocystis Infections; Colorectal Neoplasms; Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — fecal specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: RFLP analysis of SSU rRNA — 1. Genomic DNA will be extracted from Blastocystis-positive fecal samples using a specific DNA Stool Mini Kit according to the manufacturer's instructions and will be stored at -20°C until use.
  2. PCR will be used to amplify a region of Blastocystis small subunit ribosomal RNA (SSU rRNA) gene.
  3. The amplified products for the SSU rRNA gene will be digested to determine the strain subtype of Blastocystis spp. using specific restriction enzymes.

SUMMARY:
Blastocystis is an anaerobic unicellular protozoal parasite infecting the gastrointestinal tract of humans and a wide range of animals. It is one of the most common enteric microorganisms with higher prevalence rates in developing than in developed countries. Feco-oral is the main route of transmission where low socioeconomic conditions, poor hygienic practices, close contact with animals, and drinking contaminated water act as major risk factors. Infection with Blastocystis was demonstrated in both symptomatic and asymptomatic people. For a long period, Blastocystis was considered a commensal organism with no pathogenic role, but recently, many studies linked it to different gastrointestinal symptoms such as nausea, diarrhea, and abdominal pain. Association with irritable bowel syndrome and colorectal cancer was also reported.

This study aims to:

- Identify subtypes of human Blastocystis isolates in Sohag by using RFLP-PCR and provide additional information on the molecular epidemiology of this parasite in our locality.

ELIGIBILITY:
Inclusion Criteria:

* Patients from outpatient clinics, Sohag hospitals.

Exclusion Criteria:

* Patients received antiparasitic drugs in the last two weeks

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: samples will be collected from outpatients with any age & sex groups from different locations (cities and villages).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
The number of cases with subtypes of human Blastocystis isolates in Sohag | 14 weeks following the startpoint of the study.
  by using RFLP-PCR

SECONDARY OUTCOMES:
The number of cases with Blastocystis infection is recorded. | 14 weeks following the startpoint of the study.
  By molecular examination of stool samples from 100 patients

IPD SHARING:
Plan to Share IPD: Undecided